CLINICAL TRIAL: NCT00897650
Title: Molecular Fingerprints in Lung Cancer: Predicting Tumor Response to Therapy
Brief Title: Protein and RNA Expression Patterns in Predicting Response to Treatment in Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christine Lovly, MD, PhD, Assistant Professor of Medicine and Cancer Biology, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 0547; P30CA068485 (NIH); VU-VICC-THO-0547 (Other: VICC); P50CA090949 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunohistochemistry; Blotting, Western; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung tumor tissue and blood samples will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung cancer: Patients with a diagnosis of invasive lung cancer.
  Interventions: Genetic: DNA/RNA sequencing and expression levels; Genetic: Protein expression analysis; Procedure: Lung tumor biopsy; Procedure: Blood sample

INTERVENTIONS:
Genetic: DNA/RNA sequencing and expression levels — Lung tumor tissue will be collected.
Genetic: Protein expression analysis — Lung tumor tissue will be collected.
  Other Names: Matrix-assisted laser desorption/ionization time of flight mass spectrometry (MALDI); Immunohistochemistry; Western blot; RPPA
Procedure: Lung tumor biopsy — Tissue will be collected by percutaneous fine needle aspiration, a percutaneous core biopsy, or during a medically indicated procedure during which lung tumor tissue will be removed
Procedure: Blood sample — Patients will be asked for a venous blood sample

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in genetic material (DNA and RNA) and may also identify protein expression patterns related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study evaluates changes in DNA, RNA, and proteins with the goal of predicting response to treatment in patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine protein and/or RNA expression patterns capable of predicting tumor response to therapy in tumor tissue samples from patients with lung cancer or suspected of having lung cancer.
* To characterize the genes and proteins found to be predictive of response in order to help elucidate the molecular biology underlying cancer chemosensitivity.
* To evaluate DNA mutations found within the lung cancer sample which may be predictive of response or resistance to certain therapeutic agents.

OUTLINE: Patients undergo collection of tumor tissue by percutaneous fine needle aspiration, core biopsy, thoracentesis, or during any medically indicated procedure involving removal of lung cancer tissue. Tissue samples are analyzed by a variety of techniques, including DNA sequencing, RNA sequencing and expression levels, protein assessment [by immunohistochemistry, western blot, Matrix-assisted laser desorption/ionization time of flight mass spectrometry (MALDI-MS]). The goal of these studies is to identify of gene mutations, gene expression levels, and proteins predictive of treatment response. Blood samples are also collected to obtain normal DNA for analysis.

After completion of study, patients will be followed until their death.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of suspected lung cancer or lung cancer

Exclusion criteria

* Inability to undergo therapy

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who have or may have lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2005-12; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
DNA, RNA, and Protein expression patterns and mutational analysis | After lung tumor tissue and blood collection.
  DNA, RNA, and Protein expression patterns and mutation status in lung tumor tissue that are capable of predicting tumor response to therapy

SECONDARY OUTCOMES:
Characterization of genes and proteins predictive of response to therapy | After lung tumor tissue and blood collection
  Identify genes and proteins predictive of response to therapy and that can be used to identify novel mechanisms underlying lung cancer behavior

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lovly, MD, PhD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/